CLINICAL TRIAL: NCT02404688
Title: Ethanol and Cannabinoid Effects on Simulated Driving and Related Cognition
Acronym: THC-ETOH
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1501015208
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cannabis; Alcohol Effect; Driving Under the Influence of Alcohol and Other Drugs
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active THC and Placebo Ethanol (Experimental)
  Interventions: Drug: Active delta-9-THC; Drug: Placebo
- Active THC and Active Ethanol (Experimental)
  Interventions: Drug: Active delta-9-THC; Drug: Active Ethanol
- Placebo THC and Active Ethanol (Experimental)
  Interventions: Drug: Placebo; Drug: Active Ethanol
- Placebo THC and Placebo Ethanol (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active delta-9-THC — Low dose (0.015 mg/kg = 1.05 mg in a 70 kg individual) THC, dissolved in alcohol. This dose is roughly equivalent to smoking approximately 1/4 of a marijuana cigarette, or "joint". Administered over 20 minutes.
  Arms: Active THC and Active Ethanol; Active THC and Placebo Ethanol
Drug: Placebo — Control: small amount of alcohol (quarter teaspoon), with no THC. Administered over 20 minutes.
  Arms: Placebo THC and Active Ethanol; Placebo THC and Placebo Ethanol
Drug: Active Ethanol — Target BrAC of 0.04% reached over 20 minutes and then clamped to maintain this dose for an additional 60 minutes. This dose is equivalent to consuming approximately 2 drinks over 1 hour. Administered over a total of 80 minutes.
  Arms: Active THC and Active Ethanol; Placebo THC and Active Ethanol
Drug: Placebo — Control: no alcohol, administered for a total of 80 minutes.
  Arms: Active THC and Placebo Ethanol; Placebo THC and Placebo Ethanol

SUMMARY:
The overarching goal of this study is to characterize the effects of ethanol and cannabinoids on simulated driving and related cognition.

DETAILED DESCRIPTION:
To study the effects of ethanol clamped at BAC 0.04% and THC (1.05 mg in a 70 kg individual) on driving.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 21 to 55 years of age (extremes included).
* Exposed to cannabis at least once.
* Exposed to alcohol at least once.
* Able to provide informed consent.

Exclusion Criteria:

* Cannabis naive.
* Alcohol naive.
* Positive pregnancy screen
* Hearing deficits.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Road Tracking Error | baseline, +20, +50, +120, +180 mins after start of alcohol and THC infusion
  changes in road tracking errors between timepoints to assess the effects of alcohol and THC on road tracking errors.

SECONDARY OUTCOMES:
Biphasic Alcohol Effects Scale (BAES) | baseline, +20, +50, +120, +180, +240 mins after start of alcohol and THC infusion
  A scale designed to assess the stimulant and sedative effects associated with alcohol intoxication.
Visual Analog Scale (VAS) | baseline, +20, +50, +120, +180 mins after start of alcohol and THC infusion
  Feeling states associated with alcohol and cannabis intoxication will be measured using this self-report scale of feeling states.
Cognitive Test Battery | +40 mins after start of alcohol and THC infusion
  Several computer tasks will be administered to assess alcohol and THC effects on driving related cognition, including: visual vigilance, visual motor function, attention and working memory, and processing speed.
Willingness to Drive Scale | baseline, +20, +50, +120, +180 mins after start of alcohol and THC infusion
  Subjects will be asked to rate their willingness to drive at their current state in the context of various scenarios including willingness to drive from testing facility to a number of destinations that are different driving distances.
Number of Joints Scale | baseline, +20, +50, +120, +180 mins after start of alcohol and THC infusion
  Subjects will be asked to rate the number of standard joints that they believe they have been administered.
Number of Drinks Scale | baseline, +20, +50, +120, +180 mins after start of alcohol and THC infusion
  Subjects will be asked to rate the number of standard drinks that they believe they have been administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Biological Studies Unit, VA Connecticut Healthcare System, West Haven, Connecticut, United States